CLINICAL TRIAL: NCT00141453
Title: CS-866DM Phase 3 Clinical Study: A Double-Blind Controlled Trial in Patients With Diabetic Nephropathy and Overt Proteinuria Secondary to Type 2 Diabetes Mellitus
Brief Title: ORIENT: Olmesartan Reducing Incidence of End Stage Renal Disease in Diabetic Nephropathy Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Shuji Tsukiyama, Daiichi Sankyo Co., Ltd. Tokyo, Japan
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORIENT
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Diabetic Nephropathy; Type 2 Diabetes Mellitus; Proteinuria
Keywords: angiotensin II type I receptor blockers; diabetic nephropathy; end-stage renal disease; renal failure; type 2 diabetes; olmesartan medoxomil
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Proteinuria; Kidney Failure, Chronic; Renal Insufficiency | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Olmesartan medoxomil tablets 10mg to 40 mg
  Interventions: Drug: olmesartan medoxomil
- 2 (Placebo Comparator): Matching placebo tablets
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: olmesartan medoxomil — Tablets 10, 20, or 40 mg
  Arms: 1
Drug: Placebo Tablets — Matching placebo tablets
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of olmesartan versus placebo on the progression of diabetic renal disease.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of diabetic nephropathy in patients with type 2 diabetes
* albumin-to-creatinine ratio >= 300 mg/g creatinine in first morning urinalysis
* serum creatinine between 1.0 and 2.5 mg/dL in women and between 1.2 and 2.5 mg/dL in men

Exclusion Criteria:

* type 1 diabetes
* non-diabetic nephropathy
* history of myocardial infarction
* history of cardiac bypass grafting within 3 months
* history of percutaneous coronary intervention (PCI) within 6 months
* history of carotid artery or peripheral artery revascularization within 6 months
* stroke or transient ischemic attack (TIA) within 1 year
* unstable angina pectoris
* heart failure of NYHA functional classes III or IV
* rapid progression of kidney disease within 3 months
* severe orthostatic hypotension
* serum potassium level =<3.5 mEq(mmol)/L or =>5.5 mEq(mmol)L
* history of rapid elevation of the serum creatinine level after starting treatment with AII receptor antagonists or ACE inhibitors
* poor glycemic control: HbA1c level =>11%
* history of myocardial infarction (MI) or coronary artery bypass grafting (CABG) within 3 months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2003-04; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Director — R&D Division, Daiichi Sankyo Co., Ltd.
Locations (2):
- Hong Kong, China
- Tokyo, Japan

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Imai E, Haneda M, Chan JC, Yamasaki T, Kobayashi F, Ito S, Makino H. Reduction and residual proteinuria are therapeutic targets in type 2 diabetes with overt nephropathy: a post hoc analysis (ORIENT-proteinuria). Nephrol Dial Transplant. 2013 Oct;28(10):2526-34. doi: 10.1093/ndt/gft249. Epub 2013 Sep 7. PMID 24013685
- [Derived] Imai E, Chan JC, Ito S, Yamasaki T, Kobayashi F, Haneda M, Makino H; ORIENT study investigators. Effects of olmesartan on renal and cardiovascular outcomes in type 2 diabetes with overt nephropathy: a multicentre, randomised, placebo-controlled study. Diabetologia. 2011 Dec;54(12):2978-86. doi: 10.1007/s00125-011-2325-z. Epub 2011 Oct 13. PMID 21993710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population was defined by the inclusion criteria. This study was carried out at 74 centers in Japan and 3 centers in Hong Kong. After the screening visit, the patients that met inclusion and exclusion criteria were selected to participate in the study. First Patient in: 19 May 2003.
Pre-assignment Details: During 6-week screening, patients were treated with placebo and assessed for eligibility. Eligible patients were assigned to 10mg of olmesartan or placebo. 857 were screened; 577 were randomized; 566=the full analysis set (11 who completed were excluded for protocol violations). Data are based on the participants in the full analysis set.
Groups:
- Olmesartan Medoxomil: Experimental: Olmesartan medoxomil tablets 10mg to 40 mg
- Placebo Comparator: Matching placebo tablets
Period: Overall Study
Arm/Group | Olmesartan Medoxomil | Placebo Comparator
Started | 288 | 289
Completed | 282 | 284
Not Completed | 6 | 5
Not completed — Protocol Violation | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olmesartan Medoxomil | Placebo Comparator | Total
Number analyzed (Participants) | 282 | 284 | 566
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.1) | 59.2 (8.1) | 59.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 92 | 175
  Male | 199 | 192 | 391
Region of Enrollment [Number; unit: participants]
  East Asia | 282 | 284 | 566
Use of ACE inhibitors [Number; unit: participants]
  Used ACE Inhibitors | 205 | 209 | 414
  Did not use ACE Inhibitors | 77 | 75 | 152
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 77.8 (10.4) | 77.2 (10.6) | 77.5 (10.5)
HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] | 7.11 (1.20) | 7.05 (1.24) | 7.08 (1.22)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.62 (0.32) | 1.62 (0.35) | 1.62 (0.34)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 141.7 (17.0) | 140.8 (18.0) | 141.3 (17.5)
Urinary albumin:creatinine ratio [Median (Inter-Quartile Range); unit: g/g] | 1.70 [0.77 to 3.00] | 1.69 [0.87 to 3.12] | 1.69 [0.82 to 3.03]
Urinary protein: creatinine ratio [Median (Inter-Quartile Range); unit: g/g] | 2.19 [0.99 to 3.87] | 2.05 [1.10 to 3.80] | 2.12 [1.03 to 3.82]

OUTCOME MEASURES:

1. Primary Outcome: Renal Composite Outcomes
Description: first occurrence of any of the following events: Doubling of serum creatinine level; Death; End stage renal disease
Time Frame: Randomization to 5 years
Population: Full analysis set=566
Measure: Number; unit: participants
Arm/Group | Olmesartan Medoxomil | Placebo Comparator
Number analyzed (Participants) | 282 | 284
participants | 116 | 129
Statistical Analysis 1: Comparison: Olmesartan Medoxomil vs Placebo Comparator; We planned to collect 400 patients to detect 35% risk reduction for renal outcome in olmesartan group with 80% power at 2-sided .05 alpha level. The Cox regression model was applied to estimate the hazard ratios (HR)between treatment groups with 95% confidence intervals for the renal and cardiovascular composite event rate; Test type: Superiority or Other; p = 0.79, Regression, Cox; The covariates were urinary albumin:creatinine ratio and serum creatinine at baseline & regions (Japan/Hong Kong) for the renal composite event rate; Hazard Ratio (HR) = 0.97, 95% CI [0.75 to 1.24]

2. Secondary Outcome: Number of Participants Experiencing Cardiovascular Composite Outcomes
Description: Number of participants experiencing the first occurence of any of the following: Cardiovascular death; non-fatal stroke; non-fatal myocardial infarction; hospitalization for unstable angina; lower extremity amputation; coronary/carotid/peripheral revascularization.
Time Frame: Within 5 years
Population: Full analysis set=566
Measure: Number; unit: participants
Arm/Group | Olmesartan Medoxomil | Placebo Comparator
Number analyzed (Participants) | 282 | 284
participants | 40 | 53
Statistical Analysis 1: Comparison: Olmesartan Medoxomil vs Placebo Comparator; Test type: Superiority or Other; p = 0.039, Regression, Cox; Covariates baseline urinary albumin:creatinine ratio, age and history of cardiovascular disease for cardiovascular composite event rate; Hazard Ratio (HR) = 0.64, 95% CI [0.43 to 0.98]

3. Secondary Outcome: The Change in Proteinuria
Description: The median percentage change from baseline value in urinary protein:creatinine ratio
Time Frame: Randomization to 5 years
Population: Full analysis set=566
Measure: Number; unit: Median percentage change in ratio
Arm/Group | Olmesartan Medoxomil | Placebo Comparator
Number analyzed (Participants) | 282 | 284
Median percentage change in ratio
  12-week value | -19.5 | 12.6
  48-week value | -20.0 | 6.9
  144 -week value | -24.9 | 3.1

4. Secondary Outcome: Reciprocal (1/Serum Creatinine) of Serum Creatinine
Description: The amount of serum creatinine was determined by blood tests periodically during the study. The amount of creatinine is an indication of kidney function. The reciprocal of serum creatinine is used in an equation to determine the change in kidney function from baseline. The reciprocal of the serum creatinine was monitored to detect kidney function changes over duration of the study.
Time Frame: Randomization to 5 years
Population: Full analysis set=566
Measure: Median (Inter-Quartile Range); unit: dL/mg/year
Arm/Group | Olmesartan Medoxomil | Placebo Comparator
Number analyzed (Participants) | 282 | 284
dL/mg/year | -0.071 [-0.148 to -0.032] | -0.089 [-0.151 to -0.044]

ADVERSE EVENTS:
Time Frame: From baseline to up to 226 weeks
Arm/Group | Olmesartan Medoxomil | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 147/287 | 171/288
Other Adverse Events (participants affected / at risk) | 264/287 | 265/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan Medoxomil (N=287) | Placebo Comparator (N=288)
Anaemia (Blood and lymphatic system disorders) | 1 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 4
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Neprogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 25 | 35
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 2 | 2
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Antrioventricular block complete (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 6
Cardiac failure acute (Cardiac disorders) | 2 | 7
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 12 | 12
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 2
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
sick sinus syndrome (Cardiac disorders) | 1 | 1
supraventricular tachycardia (Cardiac disorders) | 0 | 1
tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
silent myocardial infarction (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 4
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
vertigo positional (Ear and labyrinth disorders) | 0 | 1
sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
angle closure glaucoma (Eye disorders) | 1 | 0
aphakia (Eye disorders) | 1 | 0
boardline glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 12 | 11
Cataract diabetic (Eye disorders) | 0 | 1
Diabetic retinal oedema (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 2 | 0
macular oedema (Eye disorders) | 1 | 1
maculopathy (Eye disorders) | 0 | 1
retinal detachment (Eye disorders) | 2 | 3
retinal hemorrhage (Eye disorders) | 0 | 1
retinal tear (Eye disorders) | 0 | 1
retinopathy proliferative (Eye disorders) | 1 | 0
vitreous haemorrhage (Eye disorders) | 7 | 8
macular hole (Eye disorders) | 0 | 1
Adominal distension (Gastrointestinal disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 0
abdominal pain lower (Gastrointestinal disorders) | 0 | 1
anal fistula (Gastrointestinal disorders) | 1 | 0
appendicitis perforated (Gastrointestinal disorders) | 1 | 0
ascites (Gastrointestinal disorders) | 1 | 1
colitis (Gastrointestinal disorders) | 1 | 0
colonic polyp (Gastrointestinal disorders) | 5 | 11
constipation (Gastrointestinal disorders) | 0 | 1
diarroea (Gastrointestinal disorders) | 0 | 3
duodenal polyp (Gastrointestinal disorders) | 1 | 0
duodenal ulcer (Gastrointestinal disorders) | 1 | 0
duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
entrocolitis (Gastrointestinal disorders) | 1 | 0
gastric ulcer (Gastrointestinal disorders) | 1 | 1
gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
gastritis (Gastrointestinal disorders) | 2 | 2
gastritis erosive (Gastrointestinal disorders) | 0 | 1
gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
haemorrhoids (Gastrointestinal disorders) | 1 | 1
inguinal hernia (Gastrointestinal disorders) | 0 | 1
intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 2
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 4 | 1
Chills (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 3
Hernia (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 0 | 3
Sudden death (General disorders) | 3 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Arthritis viral (Infections and infestations) | 0 | 1
Bartholin's abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 5 | 4
Diabetic gangrene (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 7 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
HIV infection (Infections and infestations) | 0 | 1
Infected sebaceous cyst (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 6
Nasopharyngitis (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 0 | 1
Perianal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 8
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 4
Sialoadenitis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 7 | 6
Urosepsis (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 1
Enteritis infectious (Infections and infestations) | 2 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Intraocular lens dislocation (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Medical device site reaction (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3
Arteriogram coronary (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3
Bilirubin conjugated increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood chloride decreased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 5
Blood creatinine increased (Investigations) | 12 | 15
Blood glucose decreased (Investigations) | 2 | 5
Blood glucose increased (Investigations) | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 2
Blood pressure increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 6 | 7
C-reactive protein increased (Investigations) | 3 | 3
Colonoscopy (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Glycosylated haemoglobin increased (Investigations) | 1 | 1
Haematocrit decreased (Investigations) | 2 | 4
Haemoglobin decreased (Investigations) | 3 | 5
International normalised ratio increased (Investigations) | 0 | 1
Myoglobin blood increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 2 | 4
Serum ferritin decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 2 | 1
White blood cell count increased (Investigations) | 3 | 2
Blood phosphorus increased (Investigations) | 0 | 3
Creatinine urine increased (Investigations) | 1 | 0
Sleep study (Investigations) | 5 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 1
Urine protein/creatinine ratio decreased (Investigations) | 1 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 1
Cardiac function test (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Dexamethasone suppression test positive (Investigations) | 0 | 2
Dexamethasone suppression test (Investigations) | 1 | 1
Renal function test (Investigations) | 1 | 0
Pulmonary function test abnormal (Investigations) | 1 | 0
Endoscopy large bowel (Investigations) | 1 | 0
Investigation (Investigations) | 1 | 1
Nephrological examination (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 7 | 8
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 5 | 10
Fluid retention (Metabolism and nutrition disorders) | 3 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 15
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 2 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1
Diabetic autonomic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 2 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 3
Mononeuropathy multiplex (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Dysthymic disorder (Psychiatric disorders) | 0 | 1
Psychosomatic disease (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 7 | 3
Renal failure chronic (Renal and urinary disorders) | 4 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 4 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Catheterisation cardiac (Surgical and medical procedures) | 1 | 4
Uterine prolapse repair (Surgical and medical procedures) | 1 | 0
Vitrectomy (Surgical and medical procedures) | 1 | 0
Glaucoma surgery (Surgical and medical procedures) | 1 | 0
Coronary angioplasty (Surgical and medical procedures) | 2 | 2
Continuous positive airway pressure (Surgical and medical procedures) | 1 | 1
Hospitalisation (Surgical and medical procedures) | 3 | 3
Surgical vascular shunt (Surgical and medical procedures) | 0 | 1
Elective surgery (Surgical and medical procedures) | 0 | 1
Arteriovenous shunt operation (Surgical and medical procedures) | 2 | 2
Tooth extraction (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 9 | 13
Blood pressure management (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 2 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan Medoxomil (N=287) | Placebo Comparator (N=288)
Cataract (Eye disorders) | 44 | 45
Diabetic retinopathy (Eye disorders) | 26 | 24
Vitreous haemorrhage (Eye disorders) | 12 | 16
Colonic polyp (Gastrointestinal disorders) | 9 | 17
Constipation (Gastrointestinal disorders) | 49 | 41
Diarrhoea (Gastrointestinal disorders) | 28 | 40
Gastritis (Gastrointestinal disorders) | 16 | 19
Nausea (Gastrointestinal disorders) | 15 | 12
Toothache (Gastrointestinal disorders) | 16 | 16
Chest discomfort (General disorders) | 16 | 18
Chest pain (General disorders) | 19 | 9
Malaise (General disorders) | 7 | 16
Oedema (General disorders) | 17 | 20
Oedema peripheral (General disorders) | 65 | 76
Bronchitis (Infections and infestations) | 21 | 22
Gastroenteritis (Infections and infestations) | 26 | 14
Infuenza (Infections and infestations) | 15 | 11
Nasopharyngitis (Infections and infestations) | 105 | 106
Upper respiratory tract infection (Infections and infestations) | 59 | 57
Urinary tract infection (Infections and infestations) | 19 | 17
Contusion (Injury, poisoning and procedural complications) | 25 | 16
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 13 | 15
Gout (Metabolism and nutrition disorders) | 18 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 68 | 61
Hypoglycaemia (Metabolism and nutrition disorders) | 69 | 69
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 42
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 37
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 34
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 17
Dizziness (Nervous system disorders) | 41 | 50
Dizziness postural (Nervous system disorders) | 14 | 17
Headache (Nervous system disorders) | 26 | 24
Hypoaesthesia (Nervous system disorders) | 18 | 19
Insomnia (Psychiatric disorders) | 20 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 57
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 | 15
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 37 | 23
Eczema (Skin and subcutaneous tissue disorders) | 27 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 25
Hypotension (Vascular disorders) | 15 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of Study shall not be published without prior express written consent and approval of Sponsor. Sponsor has right to change proposed publication and/or prohibit publication and Contractor must comply with requirements of Sponsor.